CLINICAL TRIAL: NCT07376863
Title: Effects of Gince Zumba and Square Stepping Exercises on Motor and Cognitive Functions in Children With Attention-Deficit/Hyperactivity Disorder
Brief Title: Impact of Structured Exercise Programs on Cognitive, Motor and Behavioral Outcomes in Children With ADHD
Acronym: ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ceylan Ekerer, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 127/64
Record Dates: First submitted 2026-01-02; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: There are 3 groups involved in the study. Each of two of the groups joined two different kinds of exercise interventions, and the control group didnt involve any regular physical activity.
Who Masked: Outcomes Assessor
Masking Description: This was a single-blind study in which outcome assessors were blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gince Zumba Group (Experimental): Participants in this arm received the Gince Zumba exercise program conducted two times per week for eight weeks
  Interventions: Other: Gince Zumba Exercise
- Square Stepping Group (Experimental): Participants in this arm received the Square Stepping exercise program conducted two times per week for eight weeks
  Interventions: Other: Square Stepping Exercise
- Control Group (No Intervention): Participants in this arm received no regular physical activity for eight weeks

INTERVENTIONS:
Other: Gince Zumba Exercise — The Gince Zumba interventions consisted of rhythm-based aerobic exercises , requiring cognitive engagement through attention, coordination, and sequencing of movements, and aiming to support cognitive functions."
  Other Names: Gince Zumba Exercises
  Arms: Gince Zumba Group
Other: Square Stepping Exercise — The Square Stepping Exercise intervention consisted of step patterns performed on a gridded mat in group sessions,, requiring cognitive engagement through visuospatial processing, attention, working memory, and sequencing of movement patterns, and aiming to support cognitive functions."
  Arms: Square Stepping Group

SUMMARY:
The purpose of this study is to investigate the effects of structured exercise interventions (Gince Zumba and Square Stepping) on cognitive, motor and behavioral functions of children diagnosed with Attention Deficit Hyperactivity Disorder (ADHD). Specifically, this study aims to:

* compare the effects of Gince Zumba and Square Stepping on motor perfoemance, including coordination and reaction time.
* examine changes in cognitive functions, particularly attention and memory functions following each exercise intervention.
* evaluate the impact of both exercise programs on behavioral symptoms and social adaptation as reported by parents
* determine whether rhytm-based exercise (Gince Zumba) or cognitively demanding stepping exercise (Square Stepping) is more effective in imroving functional outcomes in children with ADHD.

Based on these aims, the study was conducted as follows:

* Eligible participants were randomly assigned to one of the three intervention groups ( square stepping group, gince zumba group, control group)
* All participants underwent baseline assessments prior to the interventions
* Participants in the intervention groups performed assigned activities for eight weeks, while the control group did not engage in regular physical activity during the same period.
* Following the completion of the interventions, all participants underwent post-intervention assessments

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and understand Turkish language
* Use of psychostimulant medication for at least 2 months prior to enrollment

Exclusion Criteria:

* Diagnosis of intellectual disability
* Comorbidity of medical or psychiatric
* Inability to participate in physical activity

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Stroop Color Test Completion Time | Baseline and at the end of the 8-week intervention
  The Stroop Color Test is a neuropsychological assessment used to evaluate selective attention, cognitive flexibility, and inhibitory control.
  In this study, the primary outcome is the total time required to complete the interference condition of the Stroop task, measured in seconds.
  Shorter completion time indicates better attentional control and executive functioning. Measurements will be obtained before and after the 8-week exercise intervention.
Visual-Auditory Digit Span Test Total Score | Baseline and after 8 weeks
  The Visual-Auditory Digit Span Test (VADST) is a neuropsychological assessment used to evaluate short-term memory and working memory through auditory and visual digit recall tasks.
  The primary outcome measure is the total test score, expressed in points, obtained from correct responses across all subtests.
  Higher total scores indicate better memory performance and cognitive processing capacity. The assessment will be administered at baseline and after the 8-week intervention period.

SECONDARY OUTCOMES:
Blaze Pod Reaction Time Score | Baseline and after 8 weeks
  The BlazePod system is a light-based interactive training and assessment tool used to evaluate visuomotor performance.
  The secondary outcome measure is the mean reaction time, recorded in milliseconds, representing the time elapsed between the visual stimulus and the participant's motor response.
  Shorter reaction time indicates faster visuomotor processing and motor response speed. Reaction time data will be collected digitally via the BlazePod mobile application. The assessment will be conducted at baseline and after the 8-week intervention period.
Blaze Pod Number of Hits | Baseline and after 8 weeks
  The BlazePod system is a light-based interactive assessment tool used to evaluate visuomotor performance and response accuracy.
  The secondary outcome measure is the total number of correct responses (hits) recorded during the task.
  Hits represent the number of targets successfully activated within the predefined assessment duration. Higher hit counts indicate better visuomotor coordination and task performance. Performance data will be recorded digitally via the BlazePod mobile application.
  The assessment will be conducted at baseline and after the 8-week intervention period.
Blaze Pod Total Number of Errors | Baseline and after 8 weeks
  The BlazePod system is a light-based interactive assessment tool used to evaluate visuomotor performance during goal-directed motor tasks.
  The secondary outcome measure is the total error score, calculated as the sum of missed targets (miss hits) and incorrect responses (strikes) recorded during the assessment. The total error score is expressed as a numerical count.
  Lower error scores indicate better response accuracy and motor control. All performance data will be recorded digitally via the BlazePod mobile application.
  The assessment will be conducted at baseline and after the 8-week intervention period.
Conners Parent Rating Scale Total Score | Baseline and after 8 weeks
  The Conners Parent Rating Scale (CPRS) is a standardized questionnaire used to assess behavioral symptoms associated with attention-deficit/hyperactivity disorder (ADHD) in children, as reported by parents.
  The secondary outcome measure is the total score obtained from the scale, expressed in points based on parent responses to Likert-type items.
  Higher total scores indicate greater severity of ADHD-related behavioral symptoms.
  The assessment will be completed by parents at baseline and after the 8-week intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Gonca İnce, Prof., Study Chair — Cukurova University
Locations (1):
- Cukurova University, Faculty of Medicine, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported in publications will be made available upon reasonable request to the corresponding author, subject to ethical approval and a data use agreement
Supporting Information: Study Protocol
Time Frame: Beginning after publication of the primary results
Access Criteria: Data access will be provided upon reasonable request, subject to ethical approval and a data use agreement
URL: https://www.cu.edu.tr

DOCUMENTS (1):
  • Study Protocol (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT07376863/Prot_000.pdf